CLINICAL TRIAL: NCT03126552
Title: Establishing a Controlled Human Hookworm Infection Model at Leiden University Medical Center
Acronym: CHHIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Meta Roestenberg, MD, PhD, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHHIL
Record Dates: First submitted 2017-03-29; First posted 2017-04-24 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Necator Americanus Infection
Keywords: hookworm; controlled human infection model
MeSH Terms: conditions — Ancylostomiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Four healthy hookworm-naive volunteers will be infected with 50 Necator americanus L3 larvae.
  Interventions: Biological: Necator americanus L3 larvae

INTERVENTIONS:
Biological: Necator americanus L3 larvae — 50 Necator americanus L3 larvae

SUMMARY:
Four healthy hookworm-naive volunteers will be exposed to 50 L3 Necator americanus larvae once and will retain infection for up to 2 years.

DETAILED DESCRIPTION:
Four volunteers will be exposed to 50 Necator americanus L3 larvae. Volunteers will be followed on a weekly basis until week 12 after infection. If volunteers develop a patent infection, defined by detectable egg production in stool by microscopy at any timepoint within week 9 to 12, they will be scheduled to donate faeces on request.

Two years after infection or if volunteers do not excrete eggs detectable by microscopy on week 9 to 12, volunteers will be treated with a 3-day regimen of albendazole to abrogate the infection. Retreatment with albendazole will be given to volunteers who remain positive for hookworm after treatment.

Six months after the treatment, volunteers will undergo their last visit.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

1. Subject is aged ≥ 18 and ≤ 45 years.
2. Subject has adequate understanding of the procedures of the study and agrees to abide strictly thereby.
3. Subject is able to communicate well with the investigator, is available to attend all study visits.
4. Subjects are able to respond to phone or email within 24 hours during the first 12 weeks of the study.
5. Subject agrees to refrain from blood donation to Sanquin or for other purposes throughout the study period.
6. For female subjects: subject agrees to use adequate contraception and not to breastfeed for the duration of study.
7. Subject has signed informed consent

A potential subject who meets any of the following criteria will be excluded from participation in this study:

1. Any history, or evidence at screening, of clinically significant symptoms, physical signs or abnormal laboratory values suggestive of systemic conditions, such as cardiovascular, pulmonary, renal, hepatic, neurological, dermatological, endocrine, malignant, haematological, infectious, immune-deficient, psychiatric and other disorders, which could compromise the health of the volunteer during the study or interfere with the interpretation of the study results. These include, but are not limited to, any of the following:

   * history of severe asthma or other health conditions that may require future steroid use;
   * body weight <50 kg or Body Mass Index (BMI) <18.0 or >30.0 kg/m2 at screening;
   * positive HIV, HBV or HCV screening tests;
   * the use of immune modifying drugs within three months prior to study onset (inhaled and topical corticosteroids and oral anti-histamines exempted) or expected use of such during the study period;
   * having one of the following laboratory abnormalities: ferritine <10 ug/L, transferrine <2.04 g/L or Hb <7.5 mmol/L for females or <8.5 mmol/L for males.
   * history of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years;
   * any history of treatment for severe psychiatric disease by a psychiatrist in the past year;
   * history of drug or alcohol abuse interfering with normal social function in the period of one year prior to study onset.
2. Known hypersensitivity to or contra-indications for use of albendazole. Including co-medication known to interact with albendazole metabolism (e.g. carbamazepine, phenobarbital, phenytoin, cimetidine, theophylline, dexamethasone).
3. Known type 1 hypersensitivity to amphotericin B or gentamicin.
4. For female subjects: positive urine pregnancy test at screening.
5. Positive faecal PCR or Kato-Katz for hookworm at screening, any known history of hookworm infection or treatment for hookworm infection or possible exposure to hookworm in the past.
6. Being an employee or student of the department of Parasitology of the LUMC.
7. Current or past scars, tattoos, or other disruptions of skin integrity at the intended site of larval application.
8. Subjects with planned travel to hookworm-endemic areas with a stay in non-hygienic environment during this trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
Detection of hookworm eggs by faeces microscopy (Kato-Katz) at any week between week 9 to 12 post-infection. | 12 weeks
  Detection of hookworm eggs by faeces microscopy (Kato-Katz) at any week between week 9 to 12 post-infection.

SECONDARY OUTCOMES:
Number of adverse events following single exposure to hookworm larvae | 2 years
  Number of adverse events following single exposure to hookworm larvae
Humoral (antibody) and cellular immunological changes after controlled human hookworm infection | 2 years
  Humoral (antibody) and cellular immunological changes after controlled human hookworm infection
Time to positive faeces test for hookworm as defined by Kato-Katz and qPCR | 12 weeks
  Time to positive faeces test for hookworm as defined by Kato-Katz and qPCR

CONTACTS AND LOCATIONS:
Overall Officials: Meta Roestenberg, MD, PhD, Principal Investigator — LUMC
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hoogerwerf MA, Coffeng LE, Brienen EAT, Janse JJ, Langenberg MCC, Kruize YCM, Gootjes C, Manurung MD, Dekker M, Becker L, Erkens MAA, van der Beek MT, Ganesh MS, Feijt C, Winkel BMF, Westra IM, Meij P, Loukas A, Visser LG, de Vlas SJ, Yazdanbakhsh M, van Lieshout L, Roestenberg M. New Insights Into the Kinetics and Variability of Egg Excretion in Controlled Human Hookworm Infections. J Infect Dis. 2019 Aug 9;220(6):1044-1048. doi: 10.1093/infdis/jiz218. PMID 31077279